CLINICAL TRIAL: NCT03028857
Title: Double-blind Trial of Phosphatidylcholine Supplementation During Pregnancy: Impact on Attention and Social Withdrawal at 4 Years of Age
Brief Title: Choline Supplementation During Pregnancy: Impact on Attention and Social Withdrawal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-1510
Record Dates: First submitted 2017-01-13; First posted 2017-01-23 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Child Development; Prenatal Stress
MeSH Terms: interventions — Choline; Phosphatidylcholines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants will take placebo (Placebo Comparator): Participants will take placebo. Corn oil every day in place of choline
  Interventions: Drug: Placebo
- Drug: Choline (Active Comparator): Participants will take 4500 mg of phosphatidylcholine twice per day, the equivalent of approximately 1250 mg of choline per day until delivery
  Interventions: Drug: Choline

INTERVENTIONS:
Drug: Choline — Mothers are instructed to take the capsules twice a day, five 450 mg phosphatidylcholine capsules at breakfast and five phosphatidylcholine 450 mg capsules at dinner. Increased awareness into the benefits of choline by obstetricians and pregnant women, as well as our recently published results from an observational study showing a wide distribution of serum choline concentrations in pregnant women, suggest that serum choline concentration is a more apt independent variable for analyses.
  Other Names: Phosphatidylcholine
  Arms: Drug: Choline
Drug: Placebo — Mothers are instructed to take the capsules twice a day, five placebo corn oil capsules at breakfast and five placebo corn oil capsules at dinner. Increased awareness into the benefits of choline by obstetricians and pregnant women, as well as our recently published results from an observational study showing a wide distribution of serum choline concentrations in pregnant women, suggest that serum choline concentration is a more apt independent variable for analyses.
  Other Names: Corn oil every day in place of choline
  Arms: Participants will take placebo

SUMMARY:
The goal is to determine if providing a nutritional supplement, phosphatidylcholine, to pregnant women improves early brain development with improved brain-related development during the first four years of life. Participating pregnant women will receive either phosphatidylcholine or a placebo from approximately 16 weeks gestation through birth. The primary outcome is the child's behavior at four years of age as reported by the primary caregiver. Secondary outcomes include motor development, socio-emotional development, language development, and cognitive development. Potential contributors beyond the supplement, including maternal stress and placental function will also be assessed.

DETAILED DESCRIPTION:
Choline is an essential nutrient that can be found in foods, such as egg yolks, liver, and other meats. It is important for the composition and repair of normal cellular membranes, normal brain function, and normal cardiovascular function. Research has suggested that the presence of adequate amounts of choline during pregnancy and breastfeeding can help ensure healthy fetal brain development. Additionally, adequate prenatal choline levels may have long-lasting positive effects on cognitive function, including memory. However, sufficient research has not been done on the effects of choline on pregnant women and their unborn babies. This study will evaluate the safety and effectiveness of taking choline supplements during pregnancy, and whether taking choline during pregnancy will have an effect on infant development.

Participants in this double-blind study will be randomly assigned to receive either placebo or 1250 mg of choline daily throughout pregnancy, until delivery. Vital signs will be taken, potential side effects will be assessed, and study medication will be given at each visit. Blood samples will be taken at enrollment and approximately at weeks 20, 28, 32. Children will be followed and assessed until 4 years of age.

ELIGIBILITY:
Inclusion Criteria:

* General Health: Other than pregnancy related illnesses, physically healthy expectant mothers
* ages 18-45 years
* prepregnancy BMI>18 and <45

Exclusion Criteria:

* Prior history of fetal death
* Current personal history of chronic infections, including HIV
* Current personal or family history out to first degree relatives of

  1. Trimethylaminuria
  2. Homocystinuria
* Primary language other than English or Spanish
* Evidence of noncompliance

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Behavior rated on the Child Behavior Checklist. | 4 Years of age
  Our primary behavioral outcome is behavior as measured by the Child Behavior Checklist at 4 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: Camille Hoffman, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - UCHealth, Aurora, Colorado
  - Saint Joseph Hospital, Denver, Colorado

IPD SHARING:
Plan to Share IPD: Yes
A copy of the locked database with all outcome, safety, and demographic measures will be provided as a supplement to the primary publication.

REFERENCES:
- [Background] Ross RG, Hunter SK, Hoffman MC, McCarthy L, Chambers BM, Law AJ, Leonard S, Zerbe GO, Freedman R. Perinatal Phosphatidylcholine Supplementation and Early Childhood Behavior Problems: Evidence for CHRNA7 Moderation. Am J Psychiatry. 2016 May 1;173(5):509-16. doi: 10.1176/appi.ajp.2015.15091188. Epub 2015 Dec 7. PMID 26651393